CLINICAL TRIAL: NCT02230098
Title: Effects of Remote Ischemic Conditioning on Myocardial Perfusion in Humans
Acronym: CONDI-PET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Leducq Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1-10-72-124-13
Record Dates: First submitted 2013-06-10; First posted 2014-09-03 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2013-11

CONDITIONS: Ischemic Heart Disease
Keywords: remote ischemic conditioning; ischemic heart disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remote Ischemic Conditioning (Experimental): By use of short-term obstruction of the blood supply to the arm
  Interventions: Other: Remote Ischemic Conditioning
- Before Remote Ischemic Conditioning (No Intervention)

INTERVENTIONS:
Other: Remote Ischemic Conditioning
  Arms: Remote Ischemic Conditioning

SUMMARY:
Cardiovascular disease is the second leading cause of death in Denmark, and ischemic heart disease accounts for the bulk of it. The purpose of this study is to clarify whether a mechanical method of remote ischemic conditioning in the form of short-term obstruction of the blood supply to the arm, can improve the heart's blood supply in patients with ischemic heart disease. This will be attempted through experiments on patients with ischemic heart disease and experimental animal studies with simulated cardiovascular disease.

This study will help to clarify whether remote ischemic preconditioning can be used to treat patients with ischemic heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for routine myocardial Rb82-PET scanning at Dept. of Nuclear Medicine & PET center, Aarhus University Hospital, Skejby, Denmark.
* Able to understand the written patient information and to give informed consent.

Exclusion Criteria:

* Patients not undergoing Rb82-PET with adenosine stress test.
* Strenuous exercise (running, bicycling, fitness), intake of beta-blockers or alcohol intake on the day before and on the day of investigation.
* Pregnant/nursing women.
* Fertile women not using contraceptives.
* Patients in dialysis treatment.
* Other concomitant disease or treatment that according to the investigator's assessment makes the patient unsuitable for study participation.
* Known type 2 diabetes

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Changes in myocardial blood flow (MBF) | 2 hours - Measurements will be done immediately before/after intervention
  MBF before and after intervention

SECONDARY OUTCOMES:
Difference in MBF between ischemic and non-ischemic myocardial territories. | 2 hours - Measurements will be done immediately before/after intervention
Difference in MBF between patients with and without ischemic heart disease detectable by Rb82-PET. | 2 hours - Measurements will be done immediately before/after intervention
Cardioprotection by the intervention measured by an increase in myocardial salvage in isolated rabbit hearts studied in a Langendorff model. | 6 months following last patient last visit
Relation between changes in MBF and myocardial salvage in rabbit hearts | 6 months following last patient last visit
• Differences in MBF between regions supplied by coronary arteries subsequently undergoing percutaneous intervention (PCI) and regions supplied by arteries not undergoing PCI | 6 months following last patient last visit

CONTACTS AND LOCATIONS:
Overall Officials: Roni Ranghøj Nielsen, MD, PhD, Principal Investigator — Department of Cardiology, Aarhus University Hospital; Hans Erik Bøtker, Prof, MD, PhD, DMSc, Study Director — Dept. of Cardiology, Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Region Central Denmark, Denmark